CLINICAL TRIAL: NCT01421394
Title: Spinal Cord Injury Series of Tampere - Retrospective Study
Acronym: scissors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R10069
Record Dates: First submitted 2011-08-16; First posted 2011-08-22 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2011-07

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury(SCI); diffusion tensor imaging(DTI); tractography
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single group study

SUMMARY:
This prospective study will assess thoroughly functional deficits and their significance in the light of rehabilitation in spinal cord injured patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of spinal cord injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: spinal cord injured patients in "PSHP"(pirkanmaan sairaanhoitopiiri) area
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere university hospital, Tampere, Pirkanmaa, Finland